CLINICAL TRIAL: NCT04105777
Title: Open-label, Randomized, Multicenter, Phase IV Trial Comparing Parenteral Nutrition Using Eurotubes® vs. Traditional 2/3-chamber Bags in Subjects With Metastatic or Localized Solid Tumors Requiring Parenteral Nutrition - The PEKANNUSS Trial
Brief Title: Trial Comparing Parenteral Nutrition (PN) Using Eurotubes® vs. 2/3-chamber Bags in Subjects With Solid Tumors Requiring PN (PEKANNUSS)
Acronym: PEKANNUSS
Status: Terminated | Type: Observational
Why Stopped: Low recruitment
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Other Study IDs: PEKANNUSS; AIO-LQ-0119/ass (Other: AIO (Arbeitsgemeinschaft Internistische Onkologie))
Record Dates: First submitted 2019-09-11; First posted 2019-09-26 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Solid Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Standard Low Glucose Parenteral Nutrition using Eurotubes®: Patients receive standard PN reduced in glucose in Eurotubes®.
  Interventions: Device: Parenteral Nutrition Bag Eurotube
- Standard Parenteral Nutrition using Eurotubes®.: Patients receive standard PN in Eurotubes®.
  Interventions: Device: Parenteral Nutrition Bag Eurotube
- Standard Parenteral Nutrition using 2/3-chamber bags: Patients receive PN according to the routine used by the participating site.
  Interventions: Device: Parenteral Nutrition 2/3 chamber Bag

INTERVENTIONS:
Device: Parenteral Nutrition Bag Eurotube — 7-,8- or 9-chamber bags for individualized parenteral nutrition compounding.
  Groups: Standard Low Glucose Parenteral Nutrition using Eurotubes®; Standard Parenteral Nutrition using Eurotubes®.
Device: Parenteral Nutrition 2/3 chamber Bag — Premixed 2/3-chamber bags which are eventually completed with other supplements shortly before administration by infusion into the bag.
  Groups: Standard Parenteral Nutrition using 2/3-chamber bags

SUMMARY:
Patients with inoperable metastatic or localized solid tumors who have an indication for parenteral nutrition will be enrolled and receive standard parenteral nutrition according to randomization using either 2/3-chamber bags or Eurotubes®, the latter either with or without reduced glucose. The main goal of the trial is to compare the frequency of self-administered parenteral nutrition at home (autonomy rate).

DETAILED DESCRIPTION:
This is an open-label, randomized, multicenter, investigator-initiated, phase IV trial. A total number of 216 patients will be enrolled.

Patients will be stratified according to ECOG (0-1 vs. 2 vs. 3), the modified Glasgow Prognostic Score (mGPS) (0-1 vs. 2) and whether the patient receives concurrent systemic anti-tumor treatment or not.

In a first step, patients will be randomized in a 2:1 ratio to Arm A (Standard Parenteral Nutrition using Eurotubes®) or Arm B (Standard Parenteral Nutrition using 2/3-chamber bags). Patients in Arm A will be stratified again by the same criteria as listed above and randomized in a 1:1 ratio to Arm A-1 (Standard Low Glucose Parenteral Nutrition using Eurotubes®) or Arm A-2 (Standard Parenteral Nutrition using Eurotubes®). Within the study, the patient can receive PN for a maximum of 12 months after randomization as long as the PN is still indicated and deemed necessary by the investigator.

Primary objective is to compare the frequency of self-administered parenteral nutrition at home (HPN). Main secondary objectives are to compare the incidence of catheter related infections (CRI), to compare the efficacy of parenteral nutrition (PN) in terms of body weight, C-reactive protein (CRP) and albumin levels, and overall survival (OS), to compare the Quality of life (QoL) by use of a modified HPN-PROQ questionnaire, to determine the frequency and duration of visits by the nursing service and to compare specified safety parameters.

The HPN therapy plan determined at screening and any modifications and adjustments to this plan during the course of HPN treatment will be recorded.

Anti-cancer treatment at the time of screening and any changes during the course of the HPN treatment period (e.g. type of treatment) will be documented.

Monitoring of Adverse Events and medical device deficiencies will be performed at every visit. AEs will be graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.

During the study the patient will maintain a study diary to document details of the administration of the HPN. A QoL questionnaire will be completed during regular study visits until EOT.

After completion of study treatment, patients will enter the follow-up period. During this period, they will be followed approximately every 3 months for survival.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histologically confirmed metastatic or localized solid tumor. Perioperative setting of HPN is allowed if HPN is planned for a duration of ≥ 2 months
3. ECOG performance status of 0, 1, 2 or 3
4. Indication for PN (the subject needs a PN independent of the trial)
5. PN planned for 3 or more days per week
6. Negative pregnancy test in women of childbearing potential
7. Willingness to perform double-barrier contraception during study for women of childbearing potential
8. Willingness to maintain a study diary
9. Life expectancy > 3 months
10. Written informed consent

Exclusion Criteria:

1. > 4 weeks of consecutive (3 ≥ days per week) parenteral nutrition in the last 3 months prior to study enrolment
2. Participation in another interventional clinical trial that could influence the endpoints of this trial or planned participation in such a study at the same time as this study is active (participation in other trials is possible in the follow up time for OS). The study is active, if the patients receive study treatment (PN), did not discontinue the trial for other reasons, and is still within the 12 months active study period
3. Current catheter related infection at baseline
4. Pregnancy or breastfeeding
5. Known hypertriglyceridemia ≥ CTCAE grade 3
6. Unable or unwilling to provide written informed consent and to comply with the study protocol
7. Uncontrolled diabetes mellitus
8. Congestive heart failure NYHA ≥ 3
9. Renal insufficiency GFR < 30 ml/min
10. Uncontrolled infection
11. Liver insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic or localized solid tumors requiring parenteral nutrition
Sampling Method: Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
patients' autonomy | up to 1 year
  Rate of self-administered parenteral nutrition at home (autonomy rate), defined as administration without nursing service assistance, as documented within the patient's study diary and calculated as the number of patients with autonomy divided by the total number of patients in the respective arm. Autonomy - as relevant for the primary endpoint - is achieved if the patient self-administers 70% or more of her/his total administrations (Note: Help of family members or other personal caregivers accounts for self-administration).

SECONDARY OUTCOMES:
Relative weight change | up to 1 year
  Relative weight change determined at baseline and during study visits approx. every four weeks after enrolment
Relative change of albumin and CRP | up to 1 year
  Relative change of albumin and CRP levels measured at baseline and during regular study visits
Overall survival | up to 4 years
  Overall survival (OS) defined as the time from randomization to death from any cause
Incidence and severity of adverse events | up to 12 months
  incidence and severity of adverse events according to CTCAE (Common Terminology Criteria for Adverse Events) Version 5.0 criteria as assessed every 4 weeks
Patient reported outcomes - Quality of life | up to 12 months
  Quality of life as measured by a modified HPN-PROQ questionnaire at baseline, at every visit and on EOT. For different types of questions, two scales are used, one is a 7-point-scale (range 1-7) with 1 meaning "very bad", 7 "excellent" and the numbers in between the respective intermediate states. The second scale measures 10 cm. The patients will have to put a cross on the line at the place which corresponds best to their state of the past week. 0 indicates "never" or "false" and 10 "daily" or "correct".

OTHER OUTCOMES:
Catheter related infections (CRI) | up to 12 months
  Catheter related infections (CRI) defined as the presence of bacteraemia originating from the intravenous (port) catheter - Bacteraemia must be confirmed through a blood culture according to study site-specific routine, preferably through paired quantitative blood cultures or a culture of the catheter if the catheter is removed - OR any infections originating from the intravenous (port) catheter, requiring intravenous antibiotics OR infections in the intravenous (port) catheter, requiring intravenous antibiotics or antibiotics delivered to the catheter itself or catheter removal
Catheter related complications | up to 12 months
  Catheter related complications such as line occlusions of catheter-related central venous thrombosis
severe infections | up to 12 months
  Severe, NCI-CTC common toxicity criteria version 5.0 grade 3-5, infections including fever of unknown origin and other Adverse Events according to NCI-CTC common toxicity criteria version 5.0
PN-Related Adverse Events (AEs) | up to 12 months
  PN-Related Adverse Events (AEs) during therapy
hospitalizations | up to 12 months
  hospitalizations during therapy

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Goetze, Principal Investigator — KHNW Frankfurt, Germany
Locations (15):
- Germany (15):
  - Berlin Spandau Vivantes Klinikum, Berlin
  - Evangelisches Klinikum Bethel gGmbh, Bielefeld, Bielefeld
  - Augusta Kranken-Anstalt gGmbH, Bochum
  - Praxis Braunschweig, Braunschweig
  - Uniklinikum Köln, Cologne
  - Krankenhaus Nordwest, Frankfurt
  - OncoResearch Lerchenfeld GmbH, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - NCT Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Universitätsmedizin Mannheim, Mannheim
  - Klinikum Hochsauerland, Meschede
  - MVZ Onko Medical GmbH Neustadt, Neustadt am Rübenberge
  - Clinical Research Stolberg GmbH, Stolberg
  - Helios Dr. Horst Schmidt Kliniken Wiesbaden, Wiesbaden

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

REFERENCES:
- [Derived] Goetze TO, Hofheinz RD, Roetzer I, Blau W, Zander T, Luley KB, Ivanyi P, Groschek M, Kreiss-Sender J, Baur C, Wolff T, Wenning B, Behringer D, Weissinger F, Kunitz A, Tschechne B, Decker-Baumann C, Frank M, Wohn L, Riedel J, Sookthai D, Schaaf M, Al-Batran SE, Haag GM; AIO Study Group. Individually compounded multi-chamber vs. standardized parenteral nutrition bags in solid tumors-A randomized clinical trial (IKF-010). Clin Nutr ESPEN. 2025 Oct;69:106-114. doi: 10.1016/j.clnesp.2025.06.040. Epub 2025 Jun 24. PMID 40571097

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT04105777/Prot_SAP_000.pdf